CLINICAL TRIAL: NCT02972749
Title: Modifiable Factors in the Management of Glaucoma - a Randomized Controlled Trial
Brief Title: Modifiable Factors and Glaucoma - RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0127-16-WOMC
Record Dates: First submitted 2016-11-20; First posted 2016-11-23 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Intraocular Pressure
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Care Provider, Investigator

ARMS (2):
- Intervention (Experimental): Recommendations for lifestyle changes which have shown to reduce IOP. recommendations include: Moderate aerobic exercise, High fiber diet, sleeping with a head elevation and moderating caffeine intake. while continuing prescribed medical therapy.
  Interventions: Behavioral: Intervention
- Control (No Intervention): No intervention. patients are instructed to continue prescribed medical therapy.

INTERVENTIONS:
Behavioral: Intervention — Recommendations for lifestyle changes which have shown to reduce IOP. recommendations include: Moderate aerobic exercise, High fiber diet, sleeping with a head elevation and moderating caffeine intake. while continuing prescribed medical therapy.
  Arms: Intervention

SUMMARY:
There is growing awareness that environmental factors, behaviors and diet are intimately related to patient health and may play a role in the pathogenesis and progression of glaucoma. Evidence from recent years has shown that some behaviors and environmental factors can affect the intraocular pressure, the primary risk factor for glaucoma. This study aims to investigate whether simple and common lifestyle inteventions such as sleeping with a head elevation, a high fiber diet, moderate aerobic exercise and moderation in caffeine intake could affect intraocular pressure and other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with glaucoma.

Exclusion Criteria:

* Not able to attend follow-up
* Contraindication for treatment or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | Following 1 month of treatment

SECONDARY OUTCOMES:
Illness perception questionnaire results | Following 1 month of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Asaf Achiron, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- The E.Wolfson Medical Center, Holon, Israel